CLINICAL TRIAL: NCT07286019
Title: Effects of Long Duration Cycling in People With Type 1 Diabetes
Acronym: PEDAL-T1D
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat de Girona (Other)
Collaborators: University Hospital of Girona Dr. Josep Trueta (Network)
Responsible Party: Principal Investigator, Josep Vehi, Full Professor in Control and Biomedical Engineering, Universitat de Girona
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UdG-PEDAL-T1D; 2025.110 (Other: Research Ethics Committee of the University Hospital Dr. Josep Trueta of Girona)
Record Dates: First submitted 2025-11-17; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: Insulin; Exercise; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance; Motor Activity

STUDY DESIGN:
Intervention Model Description: Non-randomized parallel assignment by cohort: T1D vs non T1D
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adults with type 1 diabetes (Experimental): Adults with type 1 diabetes complete one supervised outdoor gravel cycling route of ~75 km under real-world conditions that represent moderate-intensity cycling. Intensity is not prescribed by the protocol and participants will regulate their effort themselves. Participants continue their usual insulin therapy with no protocolized insulin adjustments. A Dexcom G7 sensor is started ~4 days before the event and worn through its life to capture baseline/during/post-exercise data. Saliva and urine are collected immediately before and after the ride for omics analyses.
  Interventions: Behavioral: Prolonged moderate-intensity cycling session
- Adults without diabetes (Experimental): Adults without diabetes complete the same supervised gravel cycling route of ~75 km under real-world, moderate intensity conditions. Intensity is not prescribed by the protocol and participants will regulate their effort themselves. A Dexcom G7 sensor is started ~4 days before the event and worn through its life to capture glycemic data. Saliva and urine are collected immediately before and after the ride for omics analyses.
  Interventions: Behavioral: Prolonged moderate-intensity cycling session

INTERVENTIONS:
Behavioral: Prolonged moderate-intensity cycling session — One single outdoor gravel ride (~75km) performed at a comfortable, sustainable intensity appropriate for each participant. The protocol does not prescribe specific speed, power, or heart-rate targets. Safety monitoring and on-route support will be provided to participants.

SUMMARY:
The goal of this interventional study is to build a high quality, real world multimodal dataset that combines continuous glucose monitoring (CGM), wearable and fitness data, performance metrics, and saliva and urine omics collected during a prolonged, moderate intensity outdoor gravel-cycling session in adults with type 1 diabetes (T1D).

The main questions it aims to answer are:

* Can we collect and synchronize comprehensive CGM, physiological, performance, and omics data around a single cycling session to enable further artificial intelligence (AI) model development?
* What molecular changes in saliva and urine occur during exercise, and how do they relate to glycemic outcomes?

Participants will:

* Complete a supervised ~75 km gravel-cycling route at their own pace under real-world conditions, without protocolized therapy adjustments.
* Wear a Dexcom G7 starting ~4 days before the ride and continue through the sensor lifespan to capture CGM data.
* Provide saliva and urine immediately before and after the ride for epigenomic and proteomic analyses.

This study will generate an integrated resource that supports the development and validation of AI models for predicting glucose responses to exercise in T1D and will help guide future studies on how prolonged exercise affects glucose control.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for > 5 years.
* Age between 18-60 years.
* HbA1c ≤ 8.5%.
* Body mass index between 18 and 30 kg/m².
* Physically active (≥ 4 hours/week of exercise).
* Laboratory data and EKG without alterations of the last 12 months.
* Valid Type 2 sports medical examination, which includes a monitored stress test with continuous ECG and blood pressure monitoring, as well as an official medical certificate confirming fitness to participate in this study.
* Experience using CGM sensors and be used to self-monitor blood glucose and carbohydrate counting.

Exclusion Criteria:

* Unable to ride gravel bikes.
* Unable to use clipless pedals.
* Pregnancy and breastfeeding.
* Hypoglycemia unawareness (Clarke Test > 3).
* Severe hypoglycemia in the previous 6 monhts.
* Progressive fatal disease.
* History of drug or alcohol abuse.
* Impaired liver function.
* Clinically relevant microvascular complications (macroalbuminuria, pre-proliferative and proliferative retinopathy), cardiovascular, hepatic, neurological, endocrine or other systemic disease, apart from T1D.
* Mental conditions that prevent the subject from understanding the nature, purpose and possible consequences of the study.
* Using an experimental drug or device during the prior 30 days.

Inclusion (healthy control group): adults 18-60 years without diabetes and physically active (≥ 4 hours/week of exercise) who can provide pre/post saliva and uringe samples for omics analyses.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2025-11-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with a complete multimodal dataset collected | At visit 4 ( final follow-up), approximately 8 to 9 days after the cycling event (visit 3).
  Percentage of enrolled participants for whom all planned study data are successfully collected and available in the study database at the final follow-up visit. A complete multimodal dataset is defined as: 1) continuous monitoring data for the full wear period used in the study, 2) saliva and urine samples obtained immediately before and immediately after the cycling event (visit 3), and 3) cycling performance and physiological data (heart rate, power, GPS) recorded during the gravel cycling event (visit 3).

SECONDARY OUTCOMES:
Percentage of CGM time in glucose range 70-180 mg/dl | Baseline (days -4 to -1 before the cycling event), during the cycling event (day 0), and post-event folow up (days +1 to +5 after the cycling event).
Percentage of CGM time in hypoglycemia (<54 mg/dl) | Baseline (days -4 to -1 before the cycling event), during the cycling event (day 0), and post-event folow up (days +1 to +5 after the cycling event).
Percentage of CGM time in hyperglycemia (>250 mg/dl) | Baseline (days -4 to -1 before the cycling event), during the cycling event (day 0), and post-event folow up (days +1 to +5 after the cycling event).
Number of daily hypoglycemic events | Baseline (days -4 to -1 before the cycling event), during the cycling event (day 0), and post-event folow up (days +1 to +5 after the cycling event).
  Number of events where CGM glucose values remain below 70 mg/dl for ≥ 15 minutes. Two events are considered distinct when glucose values rise above 70 mg/dl for at least 15 minutes between them.
Median glucose concentration | Baseline (days -4 to -1 before the cycling event), during the cycling event (day 0), and post-event folow up (days +1 to +5 after the cycling event).
Daily glucose variability - Coefficient of Variation | From CGM sensor insertion through the end of the CGM monitoring period (up to approximately 10 days of wear).
  Daily glucose variability assessed as the percent coefficient of variation (CV) of CGM sensor glucose values over the CGM monitoring period.
Daily glucose variability - Interquartile range | From CGM sensor insertion through the end of the CGM monitoring period (up to approximately 10 days of wear).
  Daily glucose variability assessed as the interquartile range (IQR) of CGM sensor glucsoe values over the CGM monitoring period.
Estimated HbA1c from Glucose Management Indicator | At completion of CGM data collection at 5 days after visit 3
  Average HbA1c estimated using the Glucose Management Indicator derived from CGM data.
Continuous heart-rate profile | On the day of the gravel cycling event (day 0), from the start to the end of the cycling session.
  Instantaneous heart rate, in beats per minute, recorded continuously (1-second intervals or device default sampling rate) using a chest strap heart-rate monitor (Garmin HRM-Pro or Garmin HRM 200) from the start to the end of the gravel cycling event. The resulting hear-rate time series will be stored for later exploratory analyses.
Continuous cycling power profile | On the day of the gravel cycling event (day 0), from the start to the end of the cycling session.
  Instantaneous cycling power, in watts, recorded continuously using pedal-based power meters (Favero Assioma) throughout the gravel cycling event. The resulting power time series will be stored for later exploratory analyses, including calculation of average and maximal power, normalized power, power-zone distribution, lef/right power balance, cadence, and other derived performance metrics.
Low Blood Glucose Index (LBGI) | From CGM sensor insertion through the end of the CGM monitoring period (up to approximately 10 days of wear).
  LBGI calculated from CGM sensor glucose values over the CGM monitoring period.
High Blood Glucose Index (HBGI) | From CGM sensor insertion through the end of the CGM monitoring period (up to approximately 10 days of wear).
  HBGI calculated from CGM sensor glucose values over the CGM monitoring period.

OTHER OUTCOMES:
Number of self-reported exercise events during CGM monitoring | From CGM sensor insertion to CGM sensor removal, approximately 10 days in total.
  Number of exercise sessions recorded manually by participants during CGM monitoring using the study application or diary. Exercise events are defined as the reported period plus 2 hours after exercise. For each exercise event, CGM-based glucose metrics (e.g., median glucose, interquartile range, percentage of time in predefined glucose ranges, glucose rate of change, glucose area under the curve) and associated treatment actions (correction bolus, rescue carbohydrates intake, hypoglycemic events) will be derived for exploratory analyses. The predefined gravel cycling event is characterized in separate outcomes.
Number of self-reported meal events during CGM monitoring | From CGM sensor insertion to CGM sensor removal, approximately 10 days in total.
  Number of meal events recorded by participants during CGM monitoring using the study application or diary. Meal events are defined as the reported meal time plus 4 hours. For each meal event, CGM-based glucose metrics (e.g., median glucose, interquartile range, percentage of time in predefined glucose ranges, glucose rate of change, glcuose area under the curve, hypoglycemic events) will be derived for exploratory analyses.
Total daily insulin dose during CGM monitoring | From CGM sensor insertion to CGM sensor removal, approximately 10 days in total.
  Total insulin dose per day (U/day) during CGM monitoring, calculated as the sum of basal insulin, meal boluses, and correction boluses recorded from insulin devices and/or the study application. Summary measures (e.g., mean and variability of the total daily insulin dose and basal/bolus ratio) will be derived for exploratory analyses
Total daily carbohydrate intake during CGM monitoring | From CGM sensor insertion to CGM sensor removal, approximately 10 days in total.
  Total carbohydrate intake, in grams, per day during CGM monitoring, including meal and rescue carbohydrates, recorded using the study application or diary. Summary measures (e.g., mean daily carbohydrate intake and frequency of rescue carbohydrate use) will be derived for exploratory analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Esteve, Study Director — University Hospital of Girona Dr. Josep Trueta; Josep Vehi, Principal Investigator — Universitat de Girona; Anna Prats, Principal Investigator — Escola Universitària de la Salut i l'Esport; Aleix Beneyto, Study Director — Universitat de Girona
Locations (1):
- Modeling & Intelligent Control Engineering Laboraotry (Universitat de Girona), Girona, Girona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ENIA UdG-Dexcom Chair — https://catedradexcom.udg.edu/